CLINICAL TRIAL: NCT03414359
Title: A Randomized, Double-blind Study Comparing 3% Chloroprocaine Versus 2 % Lidocaine/ Epinephrine/ Bicarbonate/ Fentanyl for Epidural Anesthesia in Elective Cesarean Delivery
Brief Title: Comparison of Chloroprocaine vs Lidocaine for Epidural Anesthesia in Cesarean Delivery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 207313
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Surgical Anesthesia, Cesarean Section
MeSH Terms: interventions — Lidocaine; chloroprocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2% Lidocaine (Active Comparator): Group LEBF received 20 ml of 2% lidocaine (combined with the following adjuncts [0.15 ml of 0.1% epinephrine, 2 ml of 8.4% sodium bicarbonate and 2 ml of 100 mcg fentanyl
  Interventions: Drug: 2% Lidocaine
- 3% Chloroprocaine (Experimental): 20 ml of 3% chloroprocaine with 4 ml 0.9% sodium chloride
  Interventions: Drug: 3% Chloroprocaine

INTERVENTIONS:
Drug: 2% Lidocaine — 2% Lidocaine using a combined spinal-epidural (CSE)
  Other Names: Xylocaine
  Arms: 2% Lidocaine
Drug: 3% Chloroprocaine — 3% Chloroprocaine using a combined spinal-epidural (CSE)
  Other Names: Nesacaine
  Arms: 3% Chloroprocaine

SUMMARY:
Regional anesthesia is commonly used for elective and emergency cesarean delivery. It provides numerous safety advantages when compared to general anesthesia for both the mother and fetus1. Epidurals also have the added benefit of being able to provide pain relief throughout labor and in the event of cesarean delivery, epidural analgesia can be "extended" to provide surgical anesthesia. Numerous studies have been performed to assess the onset times of various local anesthetics when administered through an epidural catheter. Attempts to reduce anesthetic onset time and improve the quality of intraoperative analgesia have been attempted by using different local anesthetic solutions and by the addition of other drugs to the epidural solution (such as epinephrine, fentanyl and sodium bicarbonate).

DETAILED DESCRIPTION:
Regional anesthesia is commonly used for elective and emergency cesarean delivery. It provides numerous safety advantages when compared to general anesthesia for both the mother and fetus1. Epidurals also have the added benefit of being able to provide pain relief throughout labor and in the event of cesarean delivery, epidural analgesia can be "extended" to provide surgical anesthesia. Numerous studies have been performed to assess the onset times of various local anesthetics when administered through an epidural catheter. Attempts to reduce anesthetic onset time and improve the quality of intraoperative analgesia have been attempted by using different local anesthetic solutions and by the addition of other drugs to the epidural solution (such as epinephrine, fentanyl and sodium bicarbonate).

A recent meta-analysis concluded that the optimum local anesthetic solution for extending a labor epidural from analgesia to surgical anesthesia has yet to be determined 2. In 1994, a retrospective study compared 1.5% lidocaine/bicarbonate/epinephrine mixture to 3% chloroprocaine in parturients with pre-existing epidural catheters for urgent cesarean delivery3. It was found that the chloroprocaine group had a significantly faster onset of anesthesia compared to the lidocaine group. Both drugs provided excellent anesthesia. However a high quality study comparing 3% chloroprocaine with 2% lidocaine/ epinephrine/ bicarbonate/ fentanyl (LEBF) in terms of anesthetic onset times has yet to be performed.

Women in labor frequently request an epidural to provide pain relief. Epidural pain relief is commonly provided by the administration of a low concentration of local anesthetic and opioid solution through an epidural catheter. This solution is delivered by an automated epidural infusion pump. In the event that a cesarean delivery is required, the pre-existing epidural is frequently used to administer a higher concentration anesthetic solution to allow pain free cesarean delivery. This is commonly referred to as an "epidural top up" or as an "extension of the epidural block." Standard practice at University of Arkansas for Medical Sciences (UAMS) for an epidural top up is Lidocaine, Epinephrine, Bicarbonate and Fentanyl (LEBF) or 3% chloroprocaine. These two mixtures are routinely and almost exclusively used for epidural cesarean delivery. The decision on which mixture to use is based solely on physician preference. It is likely that the LBEF mixture is used more frequently but the investigators consider both local anesthetic mixtures as equals and the standard of care at UAMS. The investigators do not use any other local anesthetics (unless there are very specific reasons).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age for the mother
* Singleton pregnancy
* Gestation > 36 weeks
* American Society of Anesthesiologist (ASA) class II
* Provides written consent
* Infant of mother

Exclusion Criteria:

* Patient refusal
* Non-elective or urgent/emergent cesarean sections
* ASA class III or above
* Unable to understand English
* Significant back surgery or scoliosis
* Known fetal abnormality
* Weight > 120 kg
* Height < 150 cm
* Allergy to local anesthetics
* Concurrent use of sulfonamides

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Any mother requiring an elective cesarean section.
Enrollment: 70 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Sharawi, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharawi N, Bansal P, Williams M, Spencer H, Mhyre JM. Comparison of Chloroprocaine Versus Lidocaine With Epinephrine, Sodium Bicarbonate, and Fentanyl for Epidural Extension Anesthesia in Elective Cesarean Delivery: A Randomized, Triple-Blind, Noninferiority Study. Anesth Analg. 2021 Mar 1;132(3):666-675. doi: 10.1213/ANE.0000000000005141. PMID 32852294

RESULTS

PARTICIPANT FLOW:
Groups:
- 2% Lidocaine: 2% Lidocaine: 2% Lidocaine (with epinephrine, bicarbonate, and fentanyl) using a combined spinal-epidural (CSE)
Period: Overall Study
Arm/Group | 2% Lidocaine | 3% Chloroprocaine
Started | 35 | 35
Completed | 34 | 33
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2% Lidocaine | 3% Chloroprocaine | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [24 to 32] | 30 [24 to 34] | 28 [24 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 13 | 12 | 25
  Other | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 31 [27 to 37] | 32 [29 to 37] | 31 [28 to 37]
Gestational age [Median (Inter-Quartile Range); unit: days] | 273 [273 to 275] | 273 [268 to 273] | 273 [270 to 274]
Duration of epidural infusion [Median (Inter-Quartile Range); unit: minutes] | 48 [38 to 73] | 49 [36 to 70] | 49 [37 to 72]

OUTCOME MEASURES:

1. Primary Outcome: The Onset Time to Surgical Anesthesia
Description: The onset time to surgical anesthesia, as reported by the participant using a standard procedure This will be measured by the time taken from the end of the epidural loading dose to develop a loss of touch sensation using a neurotip® (Owen Mumford, USA) device bilaterally at the T7 dermatomal level using a non-inferiority study design. A non-inferiority limit of 3 minutes was chosen apriori.
Time Frame: Up to 35 minutes
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 2% Lidocaine | 3% Chloroprocaine
Number analyzed (Participants) | 34 | 33
seconds | 558 (269) | 655 (258)
Statistical Analysis 1: Comparison: 2% Lidocaine vs 3% Chloroprocaine; To exclude a clinically important difference between the LEBF group and the chloroprocaine group, given a standard deviation of 4 minutes, and a non-inferiority margin of 3 minutes difference between groups, 62 mother-infant dyads (31 mother-infant dyads in each arm) are required to have a significance level of 5% and a power of 90%. In total, 70 female patients were recruited to account for any withdrawals; Test type: Non-Inferiority — As there is no existing data in the literature that clearly defines a clinically significant reduction in the onset time of anesthesia, the non-inferiority margin was defined a priori based on clinical reasoning; p = 0.10, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is, <0.05

2. Secondary Outcome: Secondary Outcome: Number of Participants With Requirement for Intraoperative Analgesia Supplementation
Description: This requirement for any rescue medications to control discomfort or pain during CD
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | 2% Lidocaine | 3% Chloroprocaine
Number analyzed (Participants) | 34 | 33
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: During inpatient admission, approximately three days
Description: local anesthetic systemic toxicity (LAST), post-dural puncture headache (PDPH) and high spinal (defined as upper limb weakness)
Arm/Group | 2% Lidocaine | 3% Chloroprocaine
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 1/33
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2% Lidocaine (N=34) | 3% Chloroprocaine (N=33)
Post dural puncture headache (Nervous system disorders) | 0 (0) | 1 (1) — presumed post-dural puncture headache due to spinal needle, treated with epidural blood batch

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03414359/Prot_SAP_000.pdf